CLINICAL TRIAL: NCT06184464
Title: Prostatic Size Reduction Following the Administration of Leuprorelin Acetate in Localized Prostate Cancer Prior to Radiation Therapy. Pilot Study.
Brief Title: Prostatic Size Reduction Following of Leuprorelin Acetate
Acronym: PROSTSIZE
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Nicolas Feltes, M.D, Consorci Sanitari de Terrassa
Other Study IDs: PROSTATE REDUCCION
Record Dates: First submitted 2023-12-05; First posted 2023-12-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer Adenocarcinoma; Prostate Adenocarcinoma
Keywords: reduccion; Eligard; leupreline; radiotherapy; feltes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prostate patient: use of Leupreline
  Interventions: Other: ACETATE LEUPRELINE

INTERVENTIONS:
Other: ACETATE LEUPRELINE — USE ACETATE LEUPRELINE BEFORE AND AFTER PROSTATE DELIMITATION

SUMMARY:
To determine the possible reduction in prostate size following the administration of Leuprelin prior to the application of radiotherapy.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common tumor in men worldwide, including our country, with an incidence of 34,413 cases in 2020 (70.6 per 100,000 inhabitants) . The elevation of Prostate-Specific Antigen (PSA) in blood and/or an abnormality in rectal examination necessitate a prostate biopsy, the diagnostic procedure involving the extraction of a small prostate tissue sample for microscopic analysis and classification of cancer cells according to the Gleason scale (malignancy grade).

Once diagnosed, extension studies (thoraco-abdominal CT, Bone Scintigraphy, PET Choline, etc.) are conducted to rule out metastasis, the spread of tumor cells originating in the prostate, to other organs. The majority of PC cases are diagnosed at localized stages (without distant disease), allowing for local curative treatments such as surgery (Prostatectomy) and radiation therapy (Prostate Radiotherapy).

Hormonal androgen blockade (HAB) combined with radiation therapy improves oncological outcomes for localized PC . Additionally, HAB administered before radiation therapy results in a reduction in prostate gland size . This reduction allows for a decrease in the volume to be irradiated, leading to lower toxicity on surrounding healthy tissues and organs (primarily the bladder and rectum).

This apparent volume reduction is expected two months after initiating HAB, typically coinciding with the simulation CT scan for radiotherapeutic treatment planning. However, there are no studies certifying or quantifying this reduction and its subsequent benefits in PC treatment.

Currently, comparing prostate size pre- and post-HAB is challenging. The first measurement is obtained from ultrasound and/or MRI at the time of diagnosis, while the second measurement (post-HAB) is only taken during radiotherapist oncologist planning CT. This poses two problems: the inadequacy of comparing prostate sizes between different tests, and potential discrepancies in prostate delineation due to variations among different participating radiation oncologists.

ELIGIBILITY:
Inclusion Criteria:

Man with Prostate positive biopsy. Able to Ssgned informed consent form. Need of hormonal treatment before start of radiotherapy

Exclusion Criteria:

Patients With prostate size of less than 20 cc at diagnosis. Patients With Positive lymph nodes or metastatic prostate cancer disease on imaging studies.

Patients with Previous pelvic radiation therapy.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostate Cancer patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
prostate size change | at 2 months of leupreline
  comparative size between pre and post Leupreline treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided